CLINICAL TRIAL: NCT03084328
Title: Vitamin D Replacement in Nonalcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Assistant Professor, MetroHealth Medical Center
Other Study IDs: 13-00153
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients with Vitamin D level of <30ng/dL: This is a cohort of patients with fatty liver disease and also have low levels of vitamin D
  Interventions: Dietary Supplement: Vitamind D
- Patients with Vitamin D level of >30ng/dL: This is a cohort of patients with fatty liver disease and have normal levels of vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamind D — Patients will be given an over the counter vitamin D supplement of 2000 units of D3 daily for 6 months
  Groups: Patients with Vitamin D level of <30ng/dL

SUMMARY:
Vitamin D deficiency is very common in patients with fatty liver disease as evidenced by our observations in the Metabolic Liver Clinic and that reported by others. We also observed that patients with more severe fatty liver disease had lower Vitamin D concentrations. Others have shown that replacing Vitamin D in patients with cirrhosis is effective and even patients with Vitamin D replete status have lowering of Vitamin D over time if not supplemented.

One of the measures of liver injury in NAFLD is the plasma concentration of ALT and we will use this to follow patients as is currently done as standard of care. All patients in the Metabolic Liver Clinic are being routinely screened for Vitamin D deficiency as standard of care and treatment is being started with oral supplementation, but there are not standardized protocols to determine success of therapy. We hypothesize that patients with NAFLD with low Vitamin D levels will respond appropriately to Vitamin D supplementation for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults of age 18 or greater
* Diagnosis of fatty liver disease with a low Vitamin D level (< 30 ng/dl) in the past 6 months
* Able to give consent

Exclusion Criteria:

* Those currently receiving Vitamin D supplementation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population for this study is patients who have fatty liver disease. Patients who have low vitamin D (<30ng/dL) and patients who have normal vitamin D (> or = to 30ng/dL) will be followed for six months and observed.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D levels | Baseline and 6 months
  Change in plasma vitamin D levels from baseline to 6 months
Change in liver and renal function | Baseline and 6 months
  Change in hepatic function panel and renal function panel from baseline to 6 months
Change in body composition data | Baseline and 6 months
  Change in blood pressure, waist circumference, BIA and CT scan if performed clinically
Chang in lipid profile | Baseline and 6 months
  Change in HDL, LDL, and TG from baseline to 6 months
Change in insulin resistance | Basline and 6 months
  Change in insulin resistance from baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data, needs HIPPA clearance and specific IRB approval, we did not plan on original data being shared